CLINICAL TRIAL: NCT06117917
Title: Esketamine Combined With Pregabalin on Chronic Postsurgical Pain in Patients Undergoing Primary Spinal Tumor Surgery.
Brief Title: Esketamine Combined With Pregabalin on CPSP in Spinal Patients.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Smile202310
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Esketamine; Pregabaline; Chronic Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Esketamine; Pregabalin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine and pregabalin (Experimental)
  Interventions: Drug: S-ketamine and pregabalin
- Normal saline and placebo capsule (Placebo Comparator)
  Interventions: Drug: Normal saline and placebo capsule

INTERVENTIONS:
Drug: S-ketamine and pregabalin — * Drug: Pregabalin
  * 150mg (2hrs) pre operatively and 75mg twice daily post operatively for 7 days(POD1-7), followed by dose reduction to 75mg once daily for 7 days(POD8-14)
  * Drug: S-ketamine infusion
  * 0.5 mg/kg bolus after induction of anesthesia +0.12 mg/kg/h continuous intravenous infusion for 48 h
  Arms: S-ketamine and pregabalin
Drug: Normal saline and placebo capsule — * Drug: Placebo capsules
  * Two placebo capsules (2hrs) preoperatively and twice daily post operatively for 7days, followed by dose reduction to single capsule once daily for 7days
  * Drug: Normal saline
  * 0.9% saline bolus after induction of anesthesia + intravenous infusion for 48 hours
  Arms: Normal saline and placebo capsule

SUMMARY:
Chronic postsurgical pain has become one of the most common complications of surgery. The quality of life will be impacted once the postsurgical patients are combined with persistent pain. What's more, the postsurgical pain may increase other adverse outcomes. It's important to find a better way to keep the postsurgical patients away from postoperative pain. Esketamine and pregabalin have become potentially effective drugs on CPSP.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective primary spinal tumor surgery;
* Ages between 18 and 65 years old;
* American Society of Anaesthesiology (ASA) status I-III;
* Signed informed consent.

Exclusion Criteria:

* Previous adverse reaction to ketamine, s-ketamine or pregabalin;
* Patients with a diagnosed history of severe chronic pain;
* Patients with long-term analgesic treatment(gabapentin/opioids/ketamine);
* Patients with aphasia or inability to cooperate with the pain assessments;
* Known sever insufficiency of vitals(such as heart failure/renal dysfunction/hepatic failure);
* Patients with a diagnosed history of psychiatric disorder;
* Patients treated with gabapentin/pregabalin in the last three months;
* Drug abuse;
* Body mass index (BMI) > 35 kg/m2 ;
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
the proportion of patients with chronic postsurgical pain during 3 months after operation | 3 months postoperatively
  The primary outcome was the proportion of patients with CPSP during the 3-month postoperative period (defined as a NRS score ≥ 3).

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph D, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China